CLINICAL TRIAL: NCT06782867
Title: The Effect of Responsive Neurostimulation (RNS) in Treatment-resistant Obsessive-compulsive Disorder (TR-OCD)
Brief Title: RNS for Treatment-resistant Obsessive-compulsive Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNS for TR-OCD
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: OCD, RNS
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Raine syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- treatment-resistant obsessive-compulsive disorder (TR-OCD) (Experimental): Patients will undergo bilateral RNS lead implantation.
  Interventions: Device: Responsive Neurostimulation (RNS)

INTERVENTIONS:
Device: Responsive Neurostimulation (RNS) — The RNS lead is stereotactically introduced into the target in the brain and fixed to the skull; the lead is then connected to a neurostimulator implanted subcutaneously in the subclavicular region.

SUMMARY:
The purpose of this study is to investigate the effect of personalized responsive neurostimulation (RNS) therapy guided by stereoelectroencephalography (SEEG) in patients with treatment-resistant obsessive-compulsive disorder (TR-OCD).

DETAILED DESCRIPTION:
At least 40-60% of patients with obsessive-compulsive disorder (OCD) continue to have symptoms after drug treatment. There is still a lack of effective therapies for TR-OCD. In a comprehensive survey of diverse neuromodulation therapies, targeting specific nuclei with personalized responsive neurostimulation (RNS) is the most promising treatment for OCD with apparent symptoms, but the evidence remains limited. The stimulation targets of RNS for patients with TR-OCD include vALIC, BNST, amSTN, VC/VS, and NAc. The efficacy of RNS in treating OCD is closely related to precise target localization. While stereoelectroencephalography (SEEG) brain mapping can help identify Individualized effective targets and stimulation parameters. This project plans to conduct SEEG-guided RNS on TR-OCD patients to assess the safety and initial efficacy.

Another goal of this study is to examine the neuronal activity of the vALIC, BNST, amSTN, VC/VS, and NAc, respectively. At the same time, some subjects are presented with a task involving an unexpected reward and various cognitive tasks. This separate study is an option and will not affect current study participation.

Some participants will also be invited to join a related study that involves positron emission tomography (PET) scanning to determine how the stimulation changes activity in the brain. Participation in the separate PET study is optional and will not affect current study participation.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65;
2. able to provide written informed consent;
3. have a diagnosis of OCD according to the Statistical Manual of Mental Disorders-Fourth Edition-Text Revised (DSM-IV-TR) criteria and confirmed by the Mini-International Neuropsychiatric Interview Chinese version 5.0;
4. have failed to improve despite undergoing two distinct courses of selective serotonin reuptake inhibitors (SSRIs), each lasting a minimum of 3-6 months; have failed to yield therapeutic efficacy after the administration of the maximum dose of clomipramine for 3-6 months in a single trial; without achieving effectiveness under cognitive behaviour therapy for six months; have failed to achieve therapeutic efficacy after three months of atypical antipsychotic medications, singularly or in combination with SSRIs or clomipramine.

Exclusion Criteria:

1. presence of other psychotic disorders;
2. have a treatment history that includes electroconvulsive therapy (ECT), modified electroconvulsive therapy (MECT), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), DBS, and transcranial magnetic stimulation (TMS);
3. presents a suicide risk (defined as a HAMD-17 score of ≥3 on suicide-related items);
4. experience difficulty in effectively communicating with investigators;
5. with a history of traumatic brain injury (TBI);
6. with intracranial or cardiovascular stents;
7. substance abuse within the past six months;
8. unstable neurological or coagulation disorders;
9. women who are pregnant, lactating, or of childbearing potential who refuse the use of reliable contraception during the study;
10. have been involved in other clinical studies within three months before enrollment in this study;
11. any conditions unsuitable for conducting this study program considered by the study group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS): the change from baseline to 1 year in the Y-BOCS total score | 1 year
  The Y-BOCS scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms), yielding a total possible score range from 0 to 40. The total score is usually computed from the subscales for obsessions (items 1-5) and compulsions (items 6-10). The results can be interpreted based on the total score: 0-7 is sub-clinical; 8-15 is mild; 16-23 is moderate; 24-31 is severe; 32-40 is extreme.

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS): remission, response, and partial response rate | Week 2, Month 1, Month 3, Month 6, and Month 12
  remission (defined as Y-BOCS total score ≤16) at Week 2, Month 1, Month 3, Month 6, and Month 12; response is a ≥35% reduction in Y-BOCS total score from baseline to Week 2, Month 1, Month 3, Month 6, and Month 12; partial response is a 25%~34% reduction in Y-BOCS total score from baseline to Week 2, Month 1, Month 3, Month 6, and Month 12. The Y-BOCS scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms), yielding a total possible score range from 0 to 40. The total score is usually computed from the subscales for obsessions (items 1-5) and compulsions (items 6-10). The results can be interpreted based on the total score: 0-7 is sub-clinical; 8-15 is mild; 16-23 is moderate; 24-31 is severe; 32-40 is extreme.
Hamilton Anxiety Scale (HAMA): the change from baseline to 2 weeks, 1 month, 3 months, 6 months, and 1 year in the HAMA total score. | Week 2, Month 1, Month 3, Month 6, and Month 12
  HAMA is a 14-item test measuring the severity of anxiety symptoms. The total anxiety score ranges from zero to 56, with higher scores indicating more anxiety. The seven psychic anxiety items elicit a psychic anxiety score that ranges from 0 to 28. The remaining seven items yield a somatic anxiety score ranging from 0 to 28.
Hamilton Depression Rating Scale (HAMD-17): the changes of HAMD-17 scores and its subscales from baseline to 2 weeks, 1 month, 3 months, 6 months, and 1 year. | Week 2, Month 1, Month 3, Month 6, and Month 12
  HAMD-17 ranges from 0 to 52, with higher scores indicating more depression; a score of 20 or more indicates moderate to severe depression.
Pittsburgh Sleep Quality Index (PSQI): the change of PSQI from baseline to Week 2, Month 1, Month 3, Month 6, and Month 1. | Week 2, Month 1, Month 3, Month 6, and Month 12
  Consisting of 19 items, the PSQI measures several aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Clinical Global Impression-Severity (CGI-S): the change from baseline to 2 weeks, 1 month, 3 months, 6 months, and 1 year in Clinical Global Impression-Severity (CGI-S) | Week 2, Month 1, Month 3, Month 6, and Month 12
  The clinical global impression-severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. Score 1 presents normal, not at all ill, and score 7 presents among the most extremely ill patients.
Clinical Global Impression-Improvement (CGI-I): CGI-I score at Week 2, Month 1, Month 3, Month 6, and Month 12. | Week 2, Month 1, Month 3, Month 6, and Month 12
  The clinical global impression-improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Score 1 presents the patient as much improved, and score 7 presents much worse.
EuroQol-5 Dimension-level Scale (EQ-5D-5L): the change from baseline to Week 2, Month 1, Month 3, Month 6, and Month 12 in EQ-5D-5L. | Week 2, Month 1, Month 3, Month 6, and Month 12
  EQ-5D-5L is an instrument that evaluates the generic quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The score ranges from 5 (having no problems) to 25 (being unable to do/having extreme problems).
Young Mania Rating Scale (YMRS): the change from baseline to Week 2, Month 1, Month 3, Month 6, and Month 12. | Week 2, Month 1, Month 3, Month 6, and Month 12
  This scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Scores range from 0 to 60, with higher scores indicating more severe mania. A score of 0 to 5 means no obvious manic symptoms; a score of 6 to 10 means definite manic symptoms; a score of 22 or above means severe manic symptoms. It will be used as a systematic screen for DBS-induced mania or hypomania. Although scores above 8 have been considered evidence of manic symptomatology in bipolar patients, the unmasked physician will use this scale and screening questions to assess whether any hypomanic symptoms require clinical intervention including DBS adjustment.
Safety as indicated by the number of Adverse Events Week 2, Month 1, Month 3, Month 6, and Month 12. | Week 2, Month 1, Month 3, Month 6, and Month 12
  Possible Adverse Events include: Major and minor adverse events will be evaluated by Adverse Events Questionnaire (AEQ) and accompanying Case Report Form (AEQ CRF) in multiple domains, including psychiatric, neurological, and cognitive effects. The AEQ includes cognitive and behavioral screening items used in the Xuanwu DBS clinic for movement disorder patients. Additionally, we have added items for the adverse events observed in pilot DBS for OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Wang, MD & PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided